CLINICAL TRIAL: NCT05484817
Title: Early Assessment of Impaired Cardiac Function in Patients With Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician , Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: DCM2022
Record Dates: First submitted 2022-07-17; First posted 2022-08-02 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus; Left Ventricular Dysfunction
Keywords: Diabetes Mellitus; Left Ventricular Dysfunction
MeSH Terms: conditions — Diabetes Mellitus; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal cardiac function groups: Patients admitted to the hospital or recruited from the community with diabetes mellitus are screened for cardiovascular diseases by echocardiography. Global longitudinal strain (GLS) is measured by speckle tracking echocardiography. The 2015 American Society of Echocardiography guidelines recommended a mean of -20% for GLS in healthy subjects, while the upper normal limit is -18%. Therefore, the normal cardiac function groups are defined as GLS < -18%.
  Interventions: Diagnostic Test: Assessment of cardiovascular risk factor, endocrine hormones and related biomarker
- Impaired cardiac function groups: Patients admitted to the hospital or recruited from the community with diabetes mellitus are screened for cardiovascular diseases by echocardiography. Global longitudinal strain (GLS) is measured by speckle tracking echocardiography. The 2015 American Society of Echocardiography guidelines recommended a mean of -20% for GLS in healthy subjects, while the upper normal limit is -18%. Therefore, the impaired cardiac function groups are defined as GLS ≥ -18%.
  Interventions: Diagnostic Test: Assessment of cardiovascular risk factor, endocrine hormones and related biomarker

INTERVENTIONS:
Diagnostic Test: Assessment of cardiovascular risk factor, endocrine hormones and related biomarker — Cardiovascular risk factors: glycated hemoglobin/C-peptide/continuous glucose monitoring/blood pressure, blood lipids, uric acid, microalbumin test, etc. Endocrin hormones: bone metabolism, sex hormones, adrenal and pituitary hormones, and related biomarkers

SUMMARY:
This is a single-center, prospective, observational study to explore the clinical features and risk factors of impaired cardiac function detected by two-dimensional speckle tracking echocardiography in patients with diabetes mellitus. The risk factors include traditional cardiovascular risk factors, bone metabolism hormones, sex hormones, adrenal and pituitary hormones, and novel serum biomarkers.

DETAILED DESCRIPTION:
Cardiovascular complications are a leading cause of death in patients with diabetes mellitus. However, early cardiovascular disease screening presents several challenges, particularly for those who have no cardiovascular symptoms. Novel imaging techniques, such as tissue Doppler imaging and speckle tracking echocardiography, allow for the more frequent detection of early subclinical left ventricular systolic dysfunction in asymptomatic patients with diabetes. Based on speckle tracking echocardiography and other techniques, this study evaluated cardiovascular function in diabetic subjects to achieve the following objectives:

A) Investigate the clinical characteristics of diabetic patients with early cardiovascular function impairment. B) Investigate the role of traditional cardiovascular risk factors, bone metabolism hormones, sex hormones, adrenal and pituitary hormones in diabetic patients with early cardiovascular function impairment. C) Explore novel biomarkers of early cardiovascular dysfunction in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged ≥18 and ≤80 years.
2. Diagnosed type 2 or type 1 diabetes

Exclusion Criteria:

1. Moderate or severe valvular heart disease, history of thoracic surgery or congenital heart disease，atrial fibrillation.
2. History of coronary heart disease or stroke
3. Typical symptoms of cardiovascular disease（angina pectoris or limiting dyspnoea (>NYHA II)）
4. LVEF <60％
5. Malignant tumor, acute infection, abnormal liver and kidney function (ALT > normal upper limit 3 times or eGFR < 60 ml/min/1.73 m2)
6. Diabetic ketoacidosis
7. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be adults admitted to the hospital or recruited from the community with type 2 or type 1 diabetes. All patients has no medical history of known cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of impaired cardiac function in type 2 diabetes diagnosed by echocardiography | Day 1
  Proportion of participants with GLS>-18% in percent

SECONDARY OUTCOMES:
Participants' personal information by questionnaire | Day 1
  Self-reported information(history of smoking)
BMI by physical assessments | Day 1
  BMI(body mass index) in kg/m^2
Waist by physical assessments | Day 1
  Waist in kg/m^2
Systolic blood pressure by physical assessments | Day 1
  Systolic blood pressure in mmHg
Diastolic blood pressure by physical assessments | Day 1
  Diastolic blood pressure in mmHg
Glycaemic control measured by blood test | Day 1
  HbA1c in %
Fasting glucose by blood test | Day 1
  Fasting glucose in mmol/l
Islet function measured by blood test | Day 1
  Fasting C-peptide in pmol/l
Glycaemic control measured by Continuous Glucose Monitoring System | Day 1 - Day 14
  Time in range in percent
High density lipoprotein cholesterol by blood test | Day 1
  High density lipoprotein cholesterol in mmol/l
Low density lipoprotein cholesterol by blood test | Day 1
  Low density lipoprotein cholesterol in mmol/l
Total cholesterol by blood test | Day 1
  Total cholesterol in mmol/l
Triglycerides measured by blood test | Day 1
  Triglycerides in mmol/l
Masked hypertension diagnosed by ambulatory blood pressure monitoring | Day 13-Day 14
  Proportion of participants with a clinical condition in which a patient's office blood pressure (BP) level is <140/90 mm Hg but ambulatory BP readings are in the hypertensive range in percent
Uric acids measured by blood test | Day 1
  Uric acids in umol/l
Bone metabolism hormones measured by blood test | Day 1
  Osteocalcin in ng/ml
Estradiol measured by blood test | Day 1
  Estradiol in pmol/l
Testosterone measured by blood test | Day 1
  Testosterone in nmol/l
Luteinizing hormone measured by blood test | Day 1
  Luteinizing hormone in mIU/ml
Follicle-stimulating hormone measured by blood test | Day 1
  Follicle-stimulating Hormone in mIU/ml
Insulin-like growth factor 1 measured by blood test | Day 1
  Insulin-like growth factor 1 in ng/ml
Cortisol measured by blood test | Day 1
  Cortisol in nmol/l
Adrenocorticotropic-hormone measured by blood test | Day 1
  Adrenocorticotropic-hormone in pmol/l
Biomarker measured by blood test | Day 1
  Brain natriuretic peptide in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD,PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided